CLINICAL TRIAL: NCT00643617
Title: Prospective Evaluation of CyberKnife Stereotactic Radiosurgery for Low and Intermediate Risk Prostate Cancer: Emulating HDR Brachytherapy Dosimetry
Brief Title: CyberKnife Radiosurgery For Low & Intermediate Risk Prostate Cancer: Emulating HDR Brachytherapy Dosimetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accuray Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCP002.2
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer; Prostatic Cancer; Prostatic Neoplasms; Prostate Neoplasms; Cancer of the Prostate
Keywords: Prostate Cancer; CyberKnife; Stereotactic Radiosurgery; Radiosurgery; Prostate Tumor; Prostate Surgery
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Heterogeneous Dose (Other): 38 Gy delivered in 4 fractions of 9.5 Gy per fraction
  Interventions: Radiation: CyberKnife Stereotactic Radiosurgery - Low Risk; Radiation: CyberKnife Stereotactic Radiosurgery - Intermediate Risk

INTERVENTIONS:
Radiation: CyberKnife Stereotactic Radiosurgery - Low Risk — 38 Gy delivered in 4 fractions of 9.5 Gy per fraction with a radial margin of 2 mm around the prostate
  Other Names: CyberKnife
Radiation: CyberKnife Stereotactic Radiosurgery - Intermediate Risk — 38 Gy delivered in 4 fractions of 9.5 Gy per fraction with a radial margin of 5mm posterolaterally
  Other Names: CyberKnife

SUMMARY:
The purpose of this study is to investigate the effects of CyberKnife radiosurgery in patients with early stage organ-confined prostate cancer and to evaluate the effects of this treatment on the quality of life over time.

DETAILED DESCRIPTION:
In this study, CyberKnife radiosurgery will be used to produce dose distributions comparable to those created by High Dose Rate (HDR) brachytherapy treatment, without the use of invasive catheters. The radiosurgery volumes will closely be made to resemble HDR brachytherapy therapeutic volumes with similar dose limitation objectives to adjacent normal tissues.

The CyberKnife Robotic Radiosurgery System is a unique radiosurgical system capable of treating tumors anywhere in the body noninvasively and with sub-millimeter accuracy. The CyberKnife System delivers radiation using a precise targeting methodology allowing a focal treatment margin around the target, thus limiting the volume of adjacent tissue receiving high doses radiation. This in turn allows the delivery of high doses of radiation to the prostate over a short series of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Histologically proven prostate adenocarcinoma
* Biopsy within 1 year of date of registration
* Clinical Stage (CS) T1b-T2b, N0, M0
* Patients belonging to one of the following risk categories:
* Low Risk: CS T1b-T2a, Gleason Score 2-6, Prostate Specific Antigen (PSA) < or = 10 ng/ml
* Intermediate Risk: CS T2b, Gleason Score 2-6, PSA < or = 10 ng/ml or CS T1b-T2b, Gleason Score 2-6, PSA < or = 20 ng/ml or CS T1b-T2b, Gleason Score 7 and PSA < or = 10 ng/ml
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* Clinical Stage T2c or greater
* Prior prostatectomy or cryotherapy of the prostate
* Prior radiotherapy of the prostate or lower pelvis
* Implanted hardware or other material that would prohibit appropriate treatment planning or delivery
* History of an invasive malignancy other than basal or squamous skin cancers in the last 5 years
* Hormone ablation for two months prior to enrollment or during treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2007-10-22 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Fuller, MD, Study Chair — CyberKnife Centers at San Diego, CA; George Mardirossian, PhD, Study Chair — CyberKnife Centers of San Diego, CA
Locations (18):
- United States (18):
  - Mitchell Cancer Center University of South Alabama, Mobile, Alabama
  - Community Regional Medical Center, Fresno, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Pasadena Cyberknife Center, Pasadena, California
  - CyberKnife Centers of San Diego, San Diego, California
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Colorado Cyberknife, Lafayette, Colorado
  - New Millenium CyberKnife, Brandon, Florida
  - JFK Comprehensive Cancer Center, Lake Worth, Florida
  - South Florida Radiation Oncology, Wellington, Florida
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Benefis Health System - Sletten Cancer Institute, Great Falls, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - AtlantiCare Regional Medical Center, Egg Harbor, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - East Texas Medical Center, Tyler, Texas

REFERENCES:
- See also: Accuray Website — http://www.accuray.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2007 through December 2011, 307 subjects signed informed consent and were enrolled in the study at 18 centers in the United States.
Pre-assignment Details: Of these 307 subjects, 48 patients did not receive study treatment and were withdrawn from the study. Reasons for withdrawal included meeting exclusion criteria after central pathology review, insurance did not approve participation in a clinical study, or patient decision to withdraw prior to receiving treatment.
  259 subjects were assigned to either the "Low Risk" or "Intermediate Risk" groups after central pathology review results.
Groups:
- Low Risk: Patients with clinical stage (CS) Tumor (T) 1b-T2a and Gleason 2-6 and Prostate specific Antigen (PSA) ≤ 10 ng/ml
- Intermediate Risk: Patients with CS T2b and Gleason 2-6 and PSA ≤ 10 ng/ml or CS T1b-T2b and Gleason 2-6 and PSA ≤ 20 ng/ml or Gleason 7 and PSA ≤ 10 ng/ml
Period: Overall Study
Arm/Group | Low Risk | Intermediate Risk
Started (Received CyberKnife treatment) | 112 | 147
10-yr Follow up (Optional extension per protocol amendment) | 36 | 33
Completed (Completed required 5-year follow up) | 64 | 87
Not Completed | 48 | 60
Not completed — Death | 6 | 9
Not completed — Lost to Follow-up | 42 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CyberKnife Stereotactic Radiosurgery - Low Risk | CyberKnife Stereotactic Radiosurgery - Intermediate Risk | Total
Number analyzed (Participants) | 112 | 147 | 259
Age, Continuous [Mean (Full Range); unit: years] | 67.2 [45.5 to 81.9] | 68.4 [52.6 to 87.6] | 67.8 [45.5 to 87.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 112 | 147 | 259
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Black/African American | 5 | 3 | 8
  Hispanic/Latino | 1 | 12 | 13
  Native Hawaiian or Pacific Islander | 0 | 2 | 2
  White | 105 | 127 | 232
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 147 | 259
Tumor Clinical Stage (CS) [Count of Participants; unit: Participants] — Clinical T category of prostate cancer, estimated by investigator at the time of patient screening.
  Participants
    T1b = Tumor incidental histological finding in >5% of tissue resected | 0 | 0 | 0
    T1c = Tumor identified by needle biopsy found in one or both sides, but not palpable | 85 | 98 | 183
    T2a = Tumor involves ½ of one side or less | 27 | 46 | 73
    T2b = Tumor involves >½ of one side but not both sides | 0 | 3 | 3
Total Gleason Score [Count of Participants; unit: Participants] — The pathologist looking at the biopsy sample will assign one Gleason grade to the most predominant pattern in the biopsy and a second Gleason grade to the second most predominant pattern. The two grades will then be added together to determine the Gleason score. Gleason scores range from 2-10. Cancer cells that look similar to healthy cells receive a low score. Cancer cells that look less like healthy cells or look more aggressive receive a higher score.
  Patients with Gleason scores 2-6 are in the Low Risk Group. Patients with Gleason scores of 7 are in the Intermediate Risk Group.
  Participants
    Gleason 2 - 6 | 112 | 11 | 123
    Gleason 7 | 0 | 136 | 136
Prostate Specific Antigen (PSA) [Mean (Full Range); unit: ng/mL] | 4.72 [0.1 to 9.2] | 6.31 [0.9 to 19.3] | 5.6 [0.1 to 19.3]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  It was developed by the ECOG and published in 1982.
  Participants
    0 = Fully active, able to carry on all pre-disease performance without restriction | 109 | 137 | 246
    1 = Restricted in physically strenuous activity | 2 | 9 | 11
    2 = Capable of all selfcare but unable to carry out any work activities | 0 | 0 | 0
    3 = Capable of only limited selfcare | 0 | 0 | 0
    Unreported | 1 | 1 | 2
American Joint Committee on Cancer (AJCC) 6th Edition Risk Group [Count of Participants; unit: Participants]
  Low: CS T1b-T2a, Gleason 2-6, PSA ≤ 10 ng/ml | 112 | 0 | 112
  Intermediate: CS T2b, Gleason 2-6, PSA ≤ 10 ng/ml | 0 | 2 | 2
  Intermediate: CS T1b-T2b, and Gleason 2-6, PSA ≤ 20 ng/ml | 0 | 9 | 9
  Intermediate: CS T1b-T2b and Gleason 7, PSA ≤ 10 ng/ml | 0 | 136 | 136

OUTCOME MEASURES:

1. Primary Outcome: Risk for Gastrointestinal (GI) and Genitourinary (GU) Toxicity
Description: To estimate the rates of acute and late Grade 3-5 gastrointestinal and genitourinary toxicities (adverse events [AE]) observed in both low-risk and intermediate-risk cohorts during the 5 years following CyberKnife (CK) treatment for prostate cancer. Kaplan Meier estimates for 5-yr and 10-yr are reported.
  Adverse events occurring within 3 months of treatment were categorized as acute toxicities, and those developing after 3 months were considered late toxicities.
  The rates were determined using the first Grade 3 or higher adverse event per patient, reported as possibly, probably, or definitely related to CK treatment.
  The Common Toxicity Criteria for Adverse Events (CTCAE) Version 3.0 was used to determine the Grade or severity of adverse events in this study, with Grade 3 being severe or medically significant but not immediately life-threatening, Grade 4 being life-threatening and Grade 5 being death related to the adverse event.
Time Frame: Primary Safety Endpoint was measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Measure: Number; unit: percentage of participants
Groups:
- Low Risk: Patients with Clinical Stage (CS) Tumor (T)1b-T2a and Gleason 2-6 and Prostate Specific Antigen (PSA) ≤ 10 ng/ml
Arm/Group | Low Risk | Intermediate Risk
Number analyzed (Participants) | 112 | 147
percentage of participants
  Probability of experiencing Acute GI Grade 3+ event(s) | 0 | 0
  Probability of experiencing Acute GU Grade 3+ event(s) | 1.8 | 0.7
  Probability of experiencing Late GI Grade 3+ events 5 years post treatment | 0 | 0
  Probability of experiencing Late GU Grade 3+ events 5 years post treatment | 1.0 | 3.7
  Probability of experiencing Late GI Grade 3+ event(s) at 10 years post CK treatment | 0 | 0
  Probability of experiencing Late GU Grade 3+ event(s) at 10 years post CK treatment | 1.0 | 3.7

2. Primary Outcome: Biochemical Disease-Free Survival (bDFS)
Description: To determine the rate of biochemical Disease-Free Survival (bDFS), using the Phoenix definition, following CyberKnife treatment. Kaplan Meier survival curves for bDFS were created and the 5-yr and 10-yr percentages are reported.
  The Phoenix definition uses a Prostate Specific Antigen (PSA) value exceeding the patients lowest PSA value (nadir) + 2 ng/mL as an indicator of disease recurrence. The percentage of patients who did not have such a PSA rise or receive any interventional therapy to treat prostate cancer are reported below.
Time Frame: Primary Efficacy Endpoint was measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Measure: Number; unit: percentage of participants
Groups:
- Low Risk: Patients with CS T1b-T2a and Gleason 2-6 and PSA ≤ 10 ng/mL
Arm/Group | Low Risk | Intermediate Risk
Number analyzed (Participants) | 112 | 147
percentage of participants
  Probability of remaining disease-free at 5 years post-CyberKnife treatment | 100 | 89.1
  Probability of remaining disease-free at 10 years post-CyberKnife treatment | 100 | 80

3. Secondary Outcome: Disease Control and Survival Outcomes
Description: To determine the rates of local failure, distant failure, disease-free survival, disease-specific survival, and overall survival following CyberKnife treatment in prostate cancer patients.
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Measure: Number; unit: percentage of participants
Arm/Group | CyberKnife Stereotactic Radiosurgery - Low Risk | CyberKnife Stereotactic Radiosurgery - Intermediate Risk
Number analyzed (Participants) | 112 | 147
percentage of participants
  Probability of remaining free from Local Failure at 5 years post-CyberKnife treatment | 100 | 98.3
  Probability of remaining free from Local Failure at 10 years post-CyberKnife treatment | 100 | 98.3
  Probability of remaining free from Distant Failure at 5 years post-CyberKnife treatment | 100 | 95
  Probability of remaining free from Distant Failure at 10 years post-CyberKnife treatment | 100 | 95
  Probability of remaining free from disease at 5 years post-CyberKnife treatment | 100 | 89.1
  Probability of remaining free from disease at 10 years post-CyberKnife treatment | 100 | 80
  Probability of surviving prostate cancer at 5 years post-CyberKnife treatment | 100 | 100
  Probability of surviving prostate cancer at 10 years post-CyberKnife treatment | 100 | 100
  Probability of Overall survival at 5 years post-CyberKnife treatment | 95.4 | 91.7
  Probability of Overall survival at 10 years post-CyberKnife treatment | 83.8 | 86.4

4. Secondary Outcome: Quality of Life Assessments: American Urological Association (AUA) Symptom Index (SI)
Description: AUA-SI is a 7-item self-report measure used to assess urinary urgency, frequency, and voiding symptoms with scores ranging from 0 (no symptom) to 5 (symptom occurs almost always) Total score: 0-7 mild symptoms; 8-19 moderate symptoms; 20-35 severe symptoms
Time Frame: AUA questionnaire was completed at Baseline, CK Treatment, and post treatment at: 1 week, 1 month, 3 months, 6 months, and then biannually up to 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: AUA questionnaires were to be completed by patients for each follow-up visit. All questions need to be completed in order to calculate the score. During follow-up, patients may have withdrawn from the study, did not consent to continue follow-up through 10 years, were lost to follow-up, decided not to complete a questionnaire, or did not fully complete a questionnaire. Scores were calculated on fully completed questionnaires even if received/dated outside protocol specified visit window.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CyberKnife Stereotactic Radiosurgery - Low Risk: CS T1b-T2a, Gleason Score 2-6, PSA < or = 10 ng/ml
  38 Gy delivered in 4 fractions of 9.5 Gy per fraction with a radial margin of 2 mm around the prostate
- CyberKnife Stereotactic Radiosurgery - Intermediate Risk: CS T2b, Gleason Score 2-6, PSA < or = 10 ng/ml or CS T1b-T2b, Gleason Score 2-6, PSA < or = 20 ng/ml or CS T1b-T2b, Gleason Score 7 and PSA < or = 10 ng/ml
  38 Gy delivered in 4 fractions of 9.5 Gy per fraction with a radial margin of 5mm posterolaterally
Arm/Group | CyberKnife Stereotactic Radiosurgery - Low Risk | CyberKnife Stereotactic Radiosurgery - Intermediate Risk
Number analyzed (Participants) | 111 | 146
score on a scale
  Baseline: number analyzed (Participants) | 110 | 146
  Baseline | 7.05 (6.32) | 7.12 (5.79)
  Last Day of Treatment: number analyzed (Participants) | 109 | 146
  Last Day of Treatment | 9.49 (7.53) | 8.64 (7.14)
  1 Week Post Treatment: number analyzed (Participants) | 109 | 139
  1 Week Post Treatment | 13.57 (9.17) | 14.14 (8.85)
  1 Month Post Treatment: number analyzed (Participants) | 111 | 144
  1 Month Post Treatment | 11.00 (7.3) | 10.74 (6.91)
  3 Months Post Treatment: number analyzed (Participants) | 109 | 146
  3 Months Post Treatment | 7.09 (5.55) | 7.26 (5.88)
  6 Months Post Treatment: number analyzed (Participants) | 110 | 144
  6 Months Post Treatment | 7.78 (7.1) | 8.09 (6.51)
  12 Months Post Treatment: number analyzed (Participants) | 105 | 139
  12 Months Post Treatment | 8.39 (6.69) | 10.05 (7.23)
  18 Months Post Treatment: number analyzed (Participants) | 98 | 135
  18 Months Post Treatment | 8.39 (6.9) | 10.24 (8.22)
  24 Months Post Treatment: number analyzed (Participants) | 94 | 129
  24 Months Post Treatment | 7.80 (6.88) | 9.47 (7.53)
  36 Months Post Treatment: number analyzed (Participants) | 81 | 110
  36 Months Post Treatment | 7.25 (7.06) | 7.88 (6.62)
  48 Months Post Treatment: number analyzed (Participants) | 62 | 88
  48 Months Post Treatment | 6.69 (6.73) | 7.97 (6.01)
  60 Months Post Treatment: number analyzed (Participants) | 60 | 78
  60 Months Post Treatment | 7.23 (7.15) | 9.19 (7.03)
  72 Months Post Treatment: number analyzed (Participants) | 52 | 68
  72 Months Post Treatment | 7.81 (7.04) | 8.16 (7.56)
  84 Months Post Treatment: number analyzed (Participants) | 49 | 56
  84 Months Post Treatment | 7.59 (6.28) | 9.84 (8.53)
  96 Months Post Treatment: number analyzed (Participants) | 42 | 50
  96 Months Post Treatment | 8.76 (8.05) | 8.64 (6.83)
  108 Months Post Treatment: number analyzed (Participants) | 36 | 40
  108 Months Post Treatment | 8.00 (7.35) | 8.75 (6.6)
  120 Months Post Treatment: number analyzed (Participants) | 35 | 32
  120 Months Post Treatment | 7.94 (7.41) | 8.69 (6.89)

5. Secondary Outcome: Quality of Life Assessments: Expanded Prostate Cancer Index Composite (EPIC) -26 Urinary Incontinence
Description: EPIC-26 is a short form version of the Expanded Prostate Cancer Index Composite, and is a validated comprehensive instrument developed to measure the health-related quality of life among men with prostate cancer. EPIC-26 consists of 26 items under 5 domains of urinary incontinence, urinary irritative/obstructive, bowel, sexual, and hormonal.
  Answers qualitatively measure patient's bother for each symptom and are then normalized on a scale of 0 (worst) to 100 (best) to calculate domain scores if sufficient input is provided.
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: EPIC questionnaires were completed by patients at follow-up visits. A minimum number of questions needed to be completed within each domain in order to calculate a domain score. Domain scores obtained per instructions (if possible) and analyzed even if questionnaires were received/dated outside protocol specified visit window.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Low Risk: Patients with CS T1b-T2a and Gleason 2-6 and PSA ≤ 10
- Intermediate Risk: Patients with CS T2b and Gleason 2-6 and PSA ≤ 10 or CS T1b-T2b and Gleason 2-6 and PSA ≤ 20 ng/ml or Gleason 7 and PSA ≤ 10 ng/ml
Arm/Group | Low Risk | Intermediate Risk
Number analyzed (Participants) | 111 | 146
score on a scale
  Baseline | 95.77 (10.42) | 91.59 (14.39)
  1 Month Post Treatment: number analyzed (Participants) | 108 | 145
  1 Month Post Treatment | 90.33 (14.56) | 88.83 (16.85)
  6 Months Post Treatment: number analyzed (Participants) | 110 | 145
  6 Months Post Treatment | 92.81 (14.08) | 88.48 (16.51)
  12 Months Post Treatment: number analyzed (Participants) | 103 | 139
  12 Months Post Treatment | 90.64 (17.39) | 85.37 (19.23)
  24 Months Post Treatment: number analyzed (Participants) | 96 | 126
  24 Months Post Treatment | 87.66 (17.32) | 78.44 (25.72)
  36 Months Post Treatment: number analyzed (Participants) | 76 | 104
  36 Months Post Treatment | 90.2 (19.38) | 81.08 (22.8)
  48 Months Post Treatment: number analyzed (Participants) | 39 | 83
  48 Months Post Treatment | 88.74 (20.88) | 80.62 (22.11)
  60 Months Post Treatment: number analyzed (Participants) | 59 | 75
  60 Months Post Treatment | 89.5 (18.31) | 80.04 (20.8)
  72 Months Post Treatment: number analyzed (Participants) | 49 | 63
  72 Months Post Treatment | 87.44 (19.55) | 75.17 (24.86)
  84 Months Post Treatment: number analyzed (Participants) | 46 | 53
  84 Months Post Treatment | 86.26 (19.89) | 76.43 (25.68)
  96 Months Post Treatment: number analyzed (Participants) | 39 | 48
  96 Months Post Treatment | 86.32 (18.84) | 76.79 (25.46)
  108 Months Post Treatment: number analyzed (Participants) | 34 | 37
  108 Months Post Treatment | 84.17 (23.54) | 73.72 (28.88)
  120 Months Post Treatment: number analyzed (Participants) | 34 | 29
  120 Months Post Treatment | 87.04 (18.55) | 78.12 (26.25)

6. Secondary Outcome: Quality of Life Assessments: EPIC-26 Urinary Irritative Obstructive
Description: as for outcome 5
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Risk | Intermediate Risk
Number analyzed (Participants) | 111 | 146
score on a scale
  Baseline | 87.67 (13.96) | 87.59 (12.32)
  1 Month Post Treatment: number analyzed (Participants) | 108 | 145
  1 Month Post Treatment | 74.11 (17.49) | 74.03 (17.82)
  6 Months Post Treatment: number analyzed (Participants) | 110 | 145
  6 Months Post Treatment | 86.75 (14.69) | 82.91 (17.4)
  12 Months Post Treatment: number analyzed (Participants) | 103 | 139
  12 Months Post Treatment | 83.29 (15.45) | 80.1 (18.79)
  24 Months Post Treatment: number analyzed (Participants) | 96 | 126
  24 Months Post Treatment | 86.56 (15.09) | 81.05 (18.71)
  36 Months Post Treatment: number analyzed (Participants) | 76 | 104
  36 Months Post Treatment | 86.99 (15.09) | 85.77 (16.77)
  48 Months Post Treatment: number analyzed (Participants) | 39 | 83
  48 Months Post Treatment | 87.81 (13.03) | 84.03 (16.36)
  60 Months Post Treatment: number analyzed (Participants) | 59 | 75
  60 Months Post Treatment | 87.72 (14.9) | 84.15 (14.32)
  72 Months Post Treatment: number analyzed (Participants) | 49 | 63
  72 Months Post Treatment | 85.19 (13.84) | 87.95 (13.37)
  84 Months Post Treatment: number analyzed (Participants) | 46 | 53
  84 Months Post Treatment | 87.07 (13.84) | 83.13 (20.13)
  96 Months Post Treatment: number analyzed (Participants) | 39 | 48
  96 Months Post Treatment | 85.78 (14.22) | 84.58 (14.45)
  108 Months Post Treatment: number analyzed (Participants) | 34 | 37
  108 Months Post Treatment | 85.8 (14.43) | 82.09 (15.11)
  120 Months Post Treatment: number analyzed (Participants) | 34 | 29
  120 Months Post Treatment | 85.0 (17.42) | 86.25 (11.69)

7. Secondary Outcome: Quality of Life Assessments: EPIC-26 Bowel
Description: as for outcome 5
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Risk | Intermediate Risk
Number analyzed (Participants) | 111 | 146
score on a scale
  Baseline | 96.25 (8.14) | 94.84 (9.96)
  1 Month Post Treatment: number analyzed (Participants) | 108 | 145
  1 Month Post Treatment | 89.32 (14.63) | 86.05 (16.66)
  6 Months Post Treatment: number analyzed (Participants) | 110 | 145
  6 Months Post Treatment | 93.45 (12.06) | 89.92 (15.91)
  12 Months Post Treatment: number analyzed (Participants) | 103 | 139
  12 Months Post Treatment | 93.51 (11.41) | 87.97 (17.42)
  24 Months Post Treatment: number analyzed (Participants) | 96 | 126
  24 Months Post Treatment | 93.68 (11.16) | 89.28 (17.26)
  36 Months Post Treatment: number analyzed (Participants) | 76 | 104
  36 Months Post Treatment | 94.82 (9.27) | 93.29 (12.48)
  48 Months Post Treatment: number analyzed (Participants) | 39 | 83
  48 Months Post Treatment | 94.65 (9.77) | 92.04 (12.28)
  60 Months Post Treatment: number analyzed (Participants) | 59 | 75
  60 Months Post Treatment | 94.49 (11.67) | 91.03 (15.38)
  72 Months Post Treatment: number analyzed (Participants) | 49 | 63
  72 Months Post Treatment | 94.3 (10.98) | 89.54 (17.07)
  84 Months Post Treatment: number analyzed (Participants) | 46 | 53
  84 Months Post Treatment | 92.42 (11.31) | 90.49 (16.09)
  96 Months Post Treatment: number analyzed (Participants) | 39 | 48
  96 Months Post Treatment | 91.67 (14.22) | 91.27 (13.73)
  108 Months Post Treatment: number analyzed (Participants) | 34 | 37
  108 Months Post Treatment | 90.07 (12.56) | 91.33 (12.74)
  120 Months Post Treatment: number analyzed (Participants) | 34 | 29
  120 Months Post Treatment | 91.17 (13.07) | 93.59 (11.07)

8. Secondary Outcome: Quality of Life Assessments: EPIC-26 Sexual
Description: as for outcome 5
Time Frame: Secondary outcomes were measured at 5 years. Sites and patients had the option of continuing follow-up through 10 years.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Risk | Intermediate Risk
Number analyzed (Participants) | 111 | 146
score on a scale
  Baseline | 55.27 (33.41) | 56.32 (32.6)
  1 Month Post Treatment: number analyzed (Participants) | 108 | 145
  1 Month Post Treatment | 47.46 (33.58) | 50.58 (31.82)
  6 Months Post Treatment: number analyzed (Participants) | 110 | 145
  6 Months Post Treatment | 50.06 (31.91) | 51.23 (33.47)
  12 Months Post Treatment: number analyzed (Participants) | 103 | 139
  12 Months Post Treatment | 44.86 (34.82) | 45.2 (32.46)
  24 Months Post Treatment: number analyzed (Participants) | 96 | 126
  24 Months Post Treatment | 40.77 (32.15) | 39.73 (30.39)
  36 Months Post Treatment: number analyzed (Participants) | 76 | 104
  36 Months Post Treatment | 42.5 (33.57) | 40.99 (31.59)
  48 Months Post Treatment: number analyzed (Participants) | 39 | 83
  48 Months Post Treatment | 38.3 (31.56) | 38.95 (31.8)
  60 Months Post Treatment: number analyzed (Participants) | 59 | 75
  60 Months Post Treatment | 32.22 (31.16) | 36.89 (32.44)
  72 Months Post Treatment: number analyzed (Participants) | 49 | 63
  72 Months Post Treatment | 30.89 (27.26) | 33.13 (29.08)
  84 Months Post Treatment: number analyzed (Participants) | 46 | 53
  84 Months Post Treatment | 28.15 (25.51) | 35.14 (29.68)
  96 Months Post Treatment: number analyzed (Participants) | 39 | 48
  96 Months Post Treatment | 27.55 (26.55) | 34.74 (30.05)
  108 Months Post Treatment: number analyzed (Participants) | 34 | 37
  108 Months Post Treatment | 28.8 (30.09) | 36.19 (29.48)
  120 Months Post Treatment: number analyzed (Participants) | 34 | 29
  120 Months Post Treatment | 23.88 (23.55) | 33.69 (30.97)

ADVERSE EVENTS:
Time Frame: Adverse event data collected from study enrollment through end of protocol follow-up, including fiducial placement, CyberKnife radiosurgery treatment, and scheduled follow-up visits up to 10 years post-CK treatment.
Description: All adverse events were collected. Serious Adverse Events reported in clinicaltrials.gov are all events meeting serious criteria regardless of causality.
Arm/Group | Low Risk | Intermediate Risk
All-Cause Mortality (participants affected / at risk) | 9/112 | 14/147
Serious Adverse Events (participants affected / at risk) | 17/112 | 25/147
Other Adverse Events (participants affected / at risk) | 103/112 | 142/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Risk (N=112) | Intermediate Risk (N=147)
Cardiac arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Valvular Heart Disease (Cardiac disorders) | 0 (0) | 1 (1)
CNS Ischemia (Nervous system disorders) | 1 (1) | 3 (3)
Death NOS (General disorders) | 2 (2) | 4 (4)
Ischemic Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction (Small Bowel) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage/Bleeding (Gastrointestinal disorders) | 1 (1) | 2 (3)
Hemorrhage/Bleeding (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 2 (3)
Other Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (8)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cervical Spine Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mood Alteration (Nervous system disorders) | 1 (1) | 0 (0)
Transverse Myelitis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Plane crash (General disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Aortic Atheroma (Vascular disorders) | 0 (0) | 1 (1)
Kidney Transplant (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Risk (N=112) | Intermediate Risk (N=147)
Fatigue (General disorders) | 36 (38) | 36 (39)
Constipation (Gastrointestinal disorders) | 15 (15) | 18 (18)
Diarrhea (Gastrointestinal disorders) | 39 (45) | 52 (59)
Urgency (Gastrointestinal disorders) | 2 (2) | 8 (9)
Proctitis (Gastrointestinal disorders) | 8 (8) | 17 (18) — Inflammation of the rectal lining
Hemorrhage/Bleeding - GI (Gastrointestinal disorders) | 10 (10) | 18 (20) — Rectal bleeding, blood in stool
GI Pain (Gastrointestinal disorders) | 10 (11) | 21 (24) — Pain reported in the abdomen, rectum (proctalgia)
Cystitis (Renal and urinary disorders) | 9 (9) | 12 (12)
Urinary Incontinence (Renal and urinary disorders) | 12 (12) | 23 (30)
Urinary Frequency/Urgency (Renal and urinary disorders) | 75 (118) | 110 (176)
Urinary Retention (Renal and urinary disorders) | 34 (39) | 54 (65) — Hesitancy, decreased force, difficulty during urination
Hemorrhage/Bleeding - GU (Renal and urinary disorders) | 16 (19) | 36 (44) — Blood in urine (hematuria)
Urinary Tract Infection (Renal and urinary disorders) | 8 (9) | 8 (9)
Pain - GU (Renal and urinary disorders) | 59 (72) | 81 (108) — Painful urination (dysuria), pain in genitourinary region
Pain - Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (10) | 12 (14) — Pain reported in bone, joint, back, shoulder, hip
Hematospermia (Reproductive system and breast disorders) | 0 (0) | 8 (8) — Blood in sperm
Pain - Reproductive/Sexual (Reproductive system and breast disorders) | 2 (3) | 8 (10) — Pain in prostate, testes, pelvis, pain on ejaculation
Ejaculatory Dysfunction (Reproductive system and breast disorders) | 1 (1) | 7 (7)
Erectile Dysfunction (Reproductive system and breast disorders) | 26 (26) | 32 (33)

LIMITATIONS AND CAVEATS:
A limitation of this study is that of the 18 sites originally enrolling eligible patients, only 7 opted to participate in the extension of follow-up through 10 years. However, from these 7 sites, 130 patients, out of the 151 total patients who completed 5-year follow-up, consented to continue follow-up beyond 5 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT00643617/Prot_SAP_000.pdf